CLINICAL TRIAL: NCT04270344
Title: A 12-month Open-label, Multicenter Observation Study on the Occurrence of Major Adverse Cardiac Events (MACE) in Patients With Acute Myocardial Infarction (AMI) Receiving Pitavastatin/Valsartan Treatment
Brief Title: The Occurrence of MACE in Patients With AMI Receiving Pitavastatin/Valsartan Treatment
Acronym: LAMISIII
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: JW-PTVV-01
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — pitavastatin; Valsartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Pitavastatin 4mg — combination therapy with pitavastatin/valsartan (LivaloV)
  Other Names: valsartan

SUMMARY:
Prospective Observation study to identify the rate of MACE in AMI with Livalo V(Pitavastatin/Valsartan) for 12 month in Korea

DETAILED DESCRIPTION:
Following subjects with AMI event within 1 month will be assessed MACE event for 1year

* Essential hypertension or heart failure
* Idiopathic hypercholesterolemia (heterogeneous familial and non-familial hypercholesterolemia, Fredrickson classification type IIa)
* Mixed-type hypercholesterolemia (Fredrickson classification type IIb) with acute myocardial infarction (STEMI, NSTEMI),

ELIGIBILITY:
Inclusion Criteria:

* idiopathic hypercholesterolemia (heterogeneous familial and non-familial, Fredrickson type IIa) or mixed-type (Fredrickson type IIb) with AMI (STEMI, NSTEMI), including essential hypertension or heart failure
* diagnosed AMI (STEMI, NSTEMI) 1 months ago
* more than 19 years old and more than 2 years of life expectancy at screening
* informed consent

Exclusion Criteria:

* cardiogenic shock or corresponding clinical events
* contraindicated to the IP
* unsuitable to this study judged by investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: hypercholesterolemia and AMI
Sampling Method: Non-Probability Sample
Enrollment: 905 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality, non-fatal MI, repeat re-vascularization | 12 months
  MACE

SECONDARY OUTCOMES:
The rate of mortality | 6 and 12 months
  MACE
The rate of cardiac death | 6 and 12 months
  MACE
The rate of nonfatal MI | 6 and 12 months
  MACE
The rate of hospitalization due to heart failure | 6 and 12 months
  MACE
The rate of Coronary artery bypass graft(CABG) | 6 and 12 months
  MACE
The rate of target lesion re-vascularization | 6 and 12 months
  MACE
The rate of target vessel re-vascularization | 6 and 12 months
  MACE
The rate of cerebrovascular disease | 6 and 12 months
  MACE
The change of SBP, DBP | 6 and 12 months
  Hypertensive parameters
The change of TC, TG, HDL-C, LDL-C, hsCRP | 6 and 12 months
  Lipid parameters
The change of HbA1c, FBS | 6 and 12 months
  No Onset of Diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Myungho Jeong, Professor, Study Chair — Chonnam National University Hospital
Locations (1):
- JWP, Seoul, Seocho-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided